CLINICAL TRIAL: NCT05251740
Title: Impact of a Standing Program in a Child With Spina Bifida: A Case Report
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of St. Augustine for Health Sciences (Other)
Responsible Party: Principal Investigator, Marianne Hanover, PT, DPT, Physical Therapist, Principal Investigator, Assistant Professor, University of St. Augustine for Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0329-21
Record Dates: First submitted 2022-01-20; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Spina Bifida With Hydrocephalus

STUDY DESIGN:
Intervention Model Description: Single participant case study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Standing program (Experimental): The child completes a 60-minute home standing program five days per week over eight weeks.
  Interventions: Device: Altimate Medical EasyStand Bantam

INTERVENTIONS:
Device: Altimate Medical EasyStand Bantam — The child will stand in the device for 60 min per day, 5 days per week for 2 months.

SUMMARY:
The purpose of this case study is to investigate a child with MMC who has significant knee and hip flexion contractures to answer the following research questions: 1) Is a home standing program effective in reducing hip and knee flexion contractures in a child with MMC? 2) Does a home standing program result in a change in the quality of functional movement?

A Physical therapist, PT, will administer the Peds NRS and goniometric measurements prior to the start of the study and at the end of the study. The PT will also provide the parent instruction on the standing home program with weekly check-ins to ensure the parent and child are able to follow the home program. The home standing program will last 8 weeks. The parent will keep a written log of stander use. The Peds NRS scores and goniometric measurements will be compared pre and post intervention. The expected outcome is that the Peds NRS scores and hip and knee extension range of motion measurements will improve.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Spina Bifida
* be able to stand with an assistive device

Exclusion Criteria:

* a diagnosis unrelated to Spina Bifida that limits standing
* medical restrictions that contraindicate standing

Ages: 9 Years to 9 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Goniometric measurements | At 0 weeks
  A universal goniometer will be used to measure the child's hip and knee joint passive ranges of motion (PROM).
Goniometric measurements | At 8 weeks
  A universal goniometer will be used to measure the child's hip and knee joint passive ranges of motion (PROM).
Pediatric Neuromuscular Recovery Scale (Peds NRS) | At 0 weeks
  The Pediatric Neuromuscular Recovery Scale (Peds NRS) assesses the quality of functional movement in children with MMC ages 1-12years. The Peds NRS examines the quality of sitting, upper extremity function, standing, and walking.The examiner administers the Peds NRS using a height-adjustable bench, mat table, fine motor manipulatives, and a ball. The examiner scores each of the 13 items on the Peds NRS on a 12-point scale, with one point allocated to each of the 12 phases of the item. The examiner scores the highest phase achieved by the child. A summary score is obtained using the sum of the items.
Pediatric Neuromuscular Recovery Scale (Peds NRS) | At 8 weeks
  The Pediatric Neuromuscular Recovery Scale (Peds NRS) assesses the quality of functional movement in children with MMC ages 1-12years. The Peds NRS examines the quality of sitting, upper extremity function, standing, and walking.The examiner administers the Peds NRS using a height-adjustable bench, mat table, fine motor manipulatives, and a ball. The examiner scores each of the 13 items on the Peds NRS on a 12-point scale, with one point allocated to each of the 12 phases of the item. The examiner scores the highest phase achieved by the child. A summary score is obtained using the sum of the items.

CONTACTS AND LOCATIONS:
Locations (1):
- University of St. Augustine, San Marcos, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to include goniometric and Peds NRS results and describe the protocol used
Supporting Information: Study Protocol, SAP
Time Frame: July 2021, permanently